CLINICAL TRIAL: NCT01405391
Title: Phase I Multicenter, Open-label, Clinical and Pharmacokinetic Study of PM01183 on Days 1 and 8 Every Three Weeks (q3wk) in Non-Colorectal Cancer (Non-CRC) Patients
Brief Title: Study of PM01183 in Non-Colorectal Cancer Patients as a Days 1 and 8 Intravenous Short Infusion Every 3 Weeks
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-A-005-11
Record Dates: First submitted 2011-07-26; First posted 2011-07-29 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Major Advanced Solid Tumors Other Than Colorectal
Keywords: Pharma Mar; PM01183; Non-Colorectal Cancer (non-CRC); Dose finding phase I
MeSH Terms: interventions — PM 01183

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Patients will receive PM01183 on Days 1 and 8 q3wk (three weeks = one treatment cycle) as an i.v. infusion, starting at 3.0 mg/day, flat dose (FD), over a minimum total volume of 100 ml dilution (on 5% glucose or 0.9% sodium chloride) via a central catheter or over a minimum total volume of 250 ml via a peripheral line, over one hour (at a fixed rate) and through a pump device.
  Interventions: Drug: PM01183

INTERVENTIONS:
Drug: PM01183 — PM01183 drug product (DP) is presented as a lyophilized powder for concentrate for solution for infusion with two strengths, 1 mg and 4 mg vials. Before use, the 1 mg and 4 mg vials should be reconstituted with 2 ml and 8 ml of water for injection respectively, to give a solution containing 0.5 mg/ml PM01183. For administration to patients as an i.v. infusion, reconstituted vials are diluted with glucose 50 mg/ml (5%) solution for infusion or sodium chloride 9 mg/ml (0.9%) solution for infusion.

SUMMARY:
Phase I Study of PM01183 in Non-Colorectal Cancer Patients to determine the recommended dose (RD) of PM01183.

DETAILED DESCRIPTION:
Phase I Study of PM01183 in Non-Colorectal (non-CRC) Cancer Patients to determine the recommended dose (RD) of PM01183, to characterize the safety profile, compliance and feasibility of the schedule, to optimize and individualize PM01183 dosing in non-CRC patients according to individual tolerance, to characterize the pharmacokinetics (PK) of the schedule, to obtain preliminary information on the clinical antitumor activity and to perform an exploratory pharmacogenomics (PGx) analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed and dated written informed consent
2. Age ≥ 18 years.
3. Non or minimally daily activities-interfering disease related symptoms.
4. Life expectancy ≥ 3 months.
5. Patients with solid tumor other than CRC.
6. Adequate bone marrow, renal, hepatic, and metabolic function (tests within normal limits or only minimally altered as assessed ≤ 7 days before inclusion in the study)Recovery to asymptomatic or minimally altered or to baseline from any adverse event (AE) derived from previous treatment (mild alteration for alopecia, skin toxicity or fatigue are allowed).
7. Normal cardiac function cardiac function by appropriate image testing.
8. Women of childbearing potential must have a negative serum pregnancy test before study entry.

Exclusion Criteria:

1. Primary colorectal cancer diagnosis
2. Prior treatment with PM01183.
3. Concomitant diseases/conditions:

   a) History of a clinically relevant cardiac condition c) Known chronic liver disease. d) Active uncontrolled infection. e) Known human immunodeficiency virus (HIV) infection. f) Limitation of the patient's ability to comply with the treatment or follow-up protocol.
4. Symptomatic and progressive or corticosteroid-requiring documented brain metastases
5. Men or women of childbearing potential who are not using an effective method of contraception as previously described; women who are pregnant or breast feeding.
6. History of extensive prior pelvic irradiation.
7. History of previous bone marrow and/or stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Recommended dose (RD) | From treatment onset to end of treatment
  To determine the recommended dose (RD) of PM01183 administered as a 1-hour infusion intravenously (i.v.) on Days 1 and 8 every three weeks (q3wk) in non-colorectal cancer (non-CRC) patients.

SECONDARY OUTCOMES:
Pharmacokinetics (PK): The dose-exposure relationships for Cmax and area under the curve (AUC) will be evaluated. | During the infusions administered on Day 1 of Cycles 1 and 3, with a schedule of 13 samples.
  To characterize the pharmacokinetics (PK) of this schedule and explore factors that may affect individual variability in main PK parameters.
Antitumor activity measured clinically and/or radiologically according to RECIST or by evaluation of tumor markers | Every six weeks while on treatment. Patients who discontinued treatment without disease progression will be followed every three months until disease progression, other antitumor therapy, death or until the end-of-study date, whichever occurs first.
  RECIST (Response Evaluation Criteria In Solid Tumors) is a set of published rules that define when cancer patients improve ("respond"), stay the same ("stable") or worsen ("progression") during treatments.
Pharmacogenomics (PGx) analysis: Number of tumour patient samples with identified and validated putative molecular markers associated with the clinical outcome of non-CRC patients treated with PM01183. | At the end of the study (24 months)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Cancer Research Center. University of Chicago Hospitals, Chicago, Illinois

REFERENCES:
- [Derived] Fernandez-Teruel C, Lubomirov R, Fudio S. Population Pharmacokinetic-Pharmacodynamic Modeling and Covariate Analyses of Neutropenia and Thrombocytopenia in Patients With Solid Tumors Treated With Lurbinectedin. J Clin Pharmacol. 2021 Sep;61(9):1206-1219. doi: 10.1002/jcph.1886. Epub 2021 Jun 9. PMID 33914350